CLINICAL TRIAL: NCT01783522
Title: A Placebo Controlled Study to Estimate the Effect Size of Glutamine as a Supplement to Prevent Bortezomib-induced Peripheral Neuropathy in Multiple Myeloma Patients
Brief Title: Glutamine in Preventing Peripheral Neuropathy in Patients With Multiple Myeloma Receiving Bortezomib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Research Cancelled
Sponsor: Beth Faiman (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Beth Faiman, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CASE2A10; NCI-2011-01866 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-07

CONDITIONS: Chemotherapeutic Agent Toxicity; Multiple Myeloma; Peripheral Neuropathy
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (preventative nutritional supplementation) (Experimental): Patients receive glutamine PO BID. Courses repeat every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: glutamine; Other: quality-of-life assessment
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID. Courses repeat every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: quality-of-life assessment; Other: placebo

INTERVENTIONS:
Drug: glutamine — Dose of 15 grams twice times daily (to equal 30 grams a day) for a period of 4 months.
  Other Names: 2-aminoglutaramic acid; Gln; glutamic acid 5-amide; L-glutamine; NutreStore
  Arms: Arm I (preventative nutritional supplementation)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies glutamine in preventing peripheral neuropathy in patients with multiple myeloma who are receiving bortezomib. Glutamine may help prevent peripheral neuropathy in patients receiving chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the objective effect size of glutamine compared to placebo as a prophylactic intervention to prevent bortezomib-induced peripheral neuropathy in multiple myeloma patients 4 months after their first dose of study drug.

SECONDARY OBJECTIVES:

I. Estimate whether glutamine delays or prevents the onset or worsening of any neuropathy as determined by National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria.

II. Determine if glutamine may improve adherence to bortezomib therapy.

III. Assess response rate (RR) and clinical benefit response rate (CBR) according to uniform international response criteria and modified European Group for Blood and Marrow Transplantation (EBMT) criteria.

IV. Determine if glutamine may improve quality of life (QOL) at 4 months.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive glutamine orally (PO) twice daily (BID). Courses repeat every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO BID. Courses repeat every 28 days for 4 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of multiple myeloma who received bortezomib at a dose of 1.3mg/m2 SQ weekly
* No evidence of severe pre-existing peripheral neuropathy, NCI-CTCAE v4.03 =< 2
* Performance status =< 2 on the Eastern Cooperative Oncology Group (ECOG) performance scale

Exclusion Criteria:

* Concurrent use of thalidomide, vincristine, platinum compound, or other agent known to cause significant neuropathy (concurrent lenalidomide will be allowed)
* Hospitalization with clinical evidence of active infections as manifested by recurrent fevers, positive blood culture results, or requiring intravenous antibiotic therapy
* Inadequate liver and renal function with liver transaminases 3x the upper limit of normal
* Glomerular filtration rate (GFR) according to Cockcroft-Gault < 30 mL/min
* Uncontrolled congestive heart failure
* Uncontrolled mood disorders
* Fasting blood glucose >150mg/dL or blood sugar (non-fasting) >200mg/dL if no history of diabetes. Uncontrolled diabetes with HgA1C greater 7% with last evaluation.
* Seizure disorder
* Monosodium glutamate (MSG) allergy or soy allergy
* Life expectancy of shorter than 3 months based on clinical laboratory parameters and the investigator's opinion
* Uncorrected Vitamin B12 or folate deficiency on last evaluation.
* Use of over the counter (OTC) supplements other than one multivitamin tablet a day
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Faiman, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo) | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Full Range); unit: years] | 54.5 [50 to 68] | 64 [42 to 66] | 55 [42 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Degree of Peripheral Neuropathy (PNP)
Description: The Neuropathy Impairment Score -Lower Limbs (NIS-LL) is the objective measurement of PNP symptoms. The degree of PNP will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03. The CTCAE is a 0-5 scale that assesses severity of neuropathy related to cancer therapy with higher scores meaning more symptoms A difference of 2 points between groups is considered significant. This measure will be performed at baseline and at 4 months.
Time Frame: up to 4 months from start of study
Population: All participants enrolled in study and given treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Number analyzed (Participants) | 4 | 5
units on a scale | 3.40 (7.83) | 3.40 (7.83)

2. Secondary Outcome: Adherence to Bortezomib Treatment
Description: Adherence reported as a percentage based on number of doses of study drug taken divided by the expected number of doses of study drug expected to be taken for the study duration.
Time Frame: Up to 4 months
Population: All patients enrolled in study and given treatment
Measure: Number; unit: % of doses taken
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Number analyzed (Participants) | 4 | 5
% of doses taken | 100 | 98.2

3. Secondary Outcome: RR (Complete Remission [sCR+CR+Very Good Partial Remission [VGPR]+Partial Remission [PR])
Description: RR (sCR+CR+VGPR+PR) according to uniform international response criteria and CBR (RR+MR according to modified EBMT criteria) will be assessed with SPEP, 24h UPEP, serum urine immunofixation, and serum free light chain assay at the start of each cycle and after completion of the 4th cycle.
Time Frame: up to 4 months from start of study
Population: Subject data not collected due to low accrual. Research cancelled
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Average Change in Quality of Life Scores From Baseline to End of Study
Description: Quality of life will be measured on the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) including 26 summed items (responses 0 to 4 to equal a possible total score 0-108). Higher scores represent better quality of life. Average change in Quality of Life scores from baseline to end of study will be reported for each separate arm
Time Frame: from baseline to end of study at 4 months
Population: All participants enrolled in study and given treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Number analyzed (Participants) | 4 | 5
score on a scale | -7.5 (4.4) | 3.4 (11.0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 21 months
Arm/Group | Arm I (Preventative Nutritional Supplementation) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Preventative Nutritional Supplementation) (N=4) | Arm II (Placebo) (N=5)
Chills (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Preventative Nutritional Supplementation) (N=4) | Arm II (Placebo) (N=5)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (5)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (4)
Fever (General disorders) | 0 (0) | 1 (4)
Irritability (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (4)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Weight loss (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Musculoskeletal and connective tissue disorders - Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study closed early with limited accrual. Because of this, we did not collect patient data for all of the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes